CLINICAL TRIAL: NCT00237471
Title: Impact of Tight Glycaemic Control With Insulin on Novel Vascular Disease Risk Factors and Myocardial Function and Perfusion in Acute Myocardial Infarction Patients With Hyperglycaemia
Brief Title: Impact of Tight Glycaemic Control in Acute Myocardial Infarction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulty recruiting patients
Sponsor: Melbourne Health (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Dr Leo Rando, Royal Melbourne Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004.116; GEENA
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Myocardial Infarct; Hyperglycemia
Keywords: Acute Myocardial Infarction; Hyperglycaemia; Insulin Infusion
MeSH Terms: conditions — Myocardial Infarction; Hyperglycemia | interventions — Insulin

INTERVENTIONS:
Drug: Insulin (tight blood glucose control)

SUMMARY:
To determine whether tight glycaemic control with insulin improves myocardial function and myocardial perfusion (measured by myocardial contrast echocardiography) and novel vascular risk factors in patients with acute myocardial infarction and hyperglycaemia.

DETAILED DESCRIPTION:
We will randomise patients with acute myocardial infarction and blood glucose levels (BGLs) >=10mmol/L within 24 hours of pain onset, to either tight glucose control (aiming BGLs 4.5 - 7mmol/L) with an insulin infusion (for 24 hours) followed by subcutaneous insulin or standard control (BGL 6 - 12mmol/L) without the use of an insulin infusion. Serial myocardial contrast echocardiography will measure changes in myocardial perfusion and function from baseline to 3 months between each group. We will also measure changes in inflammatory and endothelial markers over this time to see whether tight glucose control improves these surrogate endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18years
* Acute Myocardial Infarction
* Blood Glucose Level >=10mmol/L
* Wall motion abnormality on baseline echocardiogram

Exclusion Criteria:

* Active infection/inflammation
* Cardiac shunt
* Cognitive Impairment
* Insulin allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-10; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Difference in the change in wall motion score index between admission, day 3-5 and after 3 months in the two treatment arms.

SECONDARY OUTCOMES:
Changes in inflammatory/endothelial markers and myocardial perfusion from admission, day 3-5 and after 3 months between the two treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Leo Rando, MBBS FRACP, Principal Investigator — Melbourne Health
Locations (1):
- The Royal Melbourne Hospital, Melbourne, Victoria, Australia